CLINICAL TRIAL: NCT05570279
Title: PLAN-A - Data- Bio-and Plan-bank Collection in Patients Treated With Radiotherapy for Squamous Cell Carcinoma of the Anus in Denmark - a DACG Cooperation
Brief Title: PLAN-A Data- Bio- and Plan- Bank Collection for SCCA in Denmark
Acronym: PLAN-A
Status: Active, not recruiting | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: Herlev Hospital (Other); Vejle Hospital (Other)
Responsible Party: Principal Investigator, Karen-Lise Garm Spindler, Professor, Aarhus University Hospital
Other Study IDs: KFE-1523
Record Dates: First submitted 2018-12-26; First posted 2022-10-06 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Anal Cancer
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue from the primary tumor and pre-treatment and consecutive blood samples are collected for a prospective biomarker evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is a prospective registration of treatment related-, toxicity-, Quality of life- and outcome data from patients treated in Denmark with radiotherapy for squamous cell carcinoma of the anus (SCCA), as a cooperation within the Danish Anal Cancer Group (DACG).

Substudy one: A prospective biobank is collected with the purpose to identify predictive and prognostic markers for outcome.

Substudy two: MRI scans are performed to investigate the rate of pelvic insufficience fractures at one year post chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Squamous cell carcinoma of the anus, and indication for curatively intended radiotherapy
* Written and oral consent

Exclusion Criteria:

* Contraindication to blood sampling or MRI scans (substudy 1 and 2)
* Other malignant disease within 5 years except from basal cell carcinomas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients eligible for radiotherapy for SCCA in Denmark will be offered inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Complete clinical response | 3 years
  Rate of complete response to primary treatment as defined by clinical and radiological evaluation

SECONDARY OUTCOMES:
Early toxicity evaluation by CTCAE | 2 weeks after the last day of therapy
  The rate of treatment related adverse events (assessed by CTCAE v.4.0) related to bowel, skin, bladder and bone.
Late toxicity evaluation by CTCAE | 1 and 3 years post treatment
  The rate of treatment related adverse events (assessed by CTCAE v.4.0) related to bowel, skin, bladder and bone.
Quality of life assessed by the EORTC QoL questionaires | 2 weeks, 1 and 3 years post therapy
  European Organisation for Research and Treatment of Cancer (EORTC) quality of life (QoL) questionnaire (QLQ) C30 (core).
  The EORTC QLQ-CR29 is a tumor-specific health related QoL questionnaire module for CRC (colorectal cancer) patients, which is designed to complement the EORTC QLQ-C30 questionnaire.
  Patients are asked to indicate their symptoms during the past week(s). Scores can be linearly transformed to provide a score from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms on the symptom scales.
Prognostic value of ctDNA | At time of treatment completion, an average of 30 days, 1 and 3 years post therapy
  Measurement of circulating tumor DNA (in copies per ML)
Incidence of pelvis fractures | 1 and 3 years post therapy
  Frequency of pelvic insufficience fractures at MRI scans

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Herlev Hospital, Herlev
  - Vejle Hospital, Vejle